CLINICAL TRIAL: NCT03495934
Title: An Open Label, Single-dose, Single-period Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Metabolite Identification of [14C]-Pracinostat in Healthy Male Subjects
Brief Title: A Study In Healthy Male Volunteers Designed To Investigate How A Radiolabelled Medicine Is Broken Down And Removed From The Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRAN-17-17
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — SB939 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single oral administration of 14C-pracinostat in the fas (Experimental)
  Interventions: Drug: pracinostat

INTERVENTIONS:
Drug: pracinostat — [14C]-pracinostat

SUMMARY:
The current study is designed to generate data for the investigation of absorption, distribution, metabolism and elimination (ADME) processes of pracinostat in humans, as well as generating samples for metabolite profiling and structural identification. The mass balance recovery of pracinostat following administration of [14C]-pracinostat will be assessed, as well as metabolite profiling and identification of pracinostat in healthy male subjects. In addition, this study will provide further PK and safety data in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. Age 40 to 65 years, inclusive
3. Body mass index of 18.0 to 35.0 kg/m2 or, if outside the range, considered not clinically significant by the investigator
4. Must be willing and able to communicate and participate in the whole study
5. Must have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day)
6. Subject is considered healthy on the basis of medical history, physical examination, triplicate electrocardiogram (ECG), vital signs and clinical laboratory assessments.
7. Provision of written informed consent to participate as shown by a signature on the volunteer consent form.
8. Male subjects must not be seeking to father a child in the next 6 months (covering 2 cycles of spermatogenesis) and must agree to use an adequate method of contraception -

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects with pregnant partners
4. Subjects who have previously been enrolled in this study
5. Subjects who have been enrolled in an absorption, distribution, metabolism and elimination (ADME) study in the last 12 months
6. History of any drug or alcohol abuse in the past 2 years
7. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit; 1.5 to 2 units = 125 mL glass of wine, depending on type)
8. Current smokers and those who have smoked within the last 12 months. A positive urine cotinine test at screening and admission
9. Current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
10. Radiation exposure, excluding background radiation but including significant medical exposures, or other trial related exposures, in the 12 months preceding participation in the trial, or radiation exposure exceeding 10 mSv in the 5 years preceding participation in the trial, inclusive of the 5 mSv exposure resulting from participation in this study. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study. Significance of a medical exposure will be determined by the investigator.
11. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening
12. Clinically significant abnormal biochemistry, haematology, coagulation or urinalysis at screening as judged by the investigator
13. Positive drugs of abuse test result
14. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
15. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <80 mL/min using the Cockcroft-Gault equation
16. Evidence of abnormal liver function at screening; alanine/aspartate aminotransferase or alkaline phosphatase > 1.5 × the upper limit of normal (ULN) or total bilirubin > 2 × ULN
17. White blood cells count (including differential), platelet count or red blood cell count below the lower limit of normal at screening
18. QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 msec (using mean of triplicate ECG)
19. History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal (GI) disease, or psychiatric disorder, as judged by the investigator
20. Subjects with a history of cholecystectomy or gall stones
21. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
22. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
23. Donation or loss of greater than 400 mL of blood within the previous 3 months
24. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the PI and sponsor's medical monitor.
25. Subjects who have used any medication, foods or lifestyle products that induces cytochrome P450 (CYP)-1A2, -2C8 or -3A4 in the past 28 days
26. Any other reason why the investigator believes participation may not be in the best interests of the potential participant -

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
mass balance recovery | up to 12 days
  urine and faeces will becollected at different time points and the radioactivity will be measured. The recovery will be expressed as percentage of radioactivity administrated
Area Under the Curve (AUC) | up to 8 days
  blood and plasma samples will be collected and the radioactivity measured to determine the Area under the concentration-time curve
Maximum concentration (Cmax) | up to 8 days
  blood and plasma samples will be collected and the radioactivity measured to determine the max concentration in concentration-time curve
clearance (CL/F) | up to 8 days
  systemic clearance after extravascular administration
Volume of distribution (Vd/F) | up to measurable concentration
  volume of distribution after extravascular administration
terminal half life (t1/2) | up to 8 days
  blood and plasma samples will be collected and the radioactivity measured to determine the terminal half life of the concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Science, Ruddington, United Kingdom